CLINICAL TRIAL: NCT01221038
Title: Preliminary Study for Standardization of Heat Tolerance Test for Young Women
Brief Title: Standardization of a Heat Tolerance Test for Young Women as a Basis for Heat Tolerance Tests in Female Soldiers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Amit Druyan, Heler Institute
Other Study IDs: 923-2010-CTIL
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-06

CONDITIONS: Heat Tolerance

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group 1: young women not using OC
- group 2: young women using OC
- group 3: young men (database)

SUMMARY:
Background:

Heat stroke is defined as a condition where the body temperature raises to dangerous level that may cause harm to body tissues and lead to multi-system clinical and pathological manifestations that might lead to death. Among heat stroke survivors a defect in thermoregulation develops as a consequence. In the IDF, every soldier who had a heat stroke, or is suspected to have had a heat stroke, must pass a heat intolerance test in the Unit of Military Physiology, after a rest period of 4-6 from the incident, which is the approximate period for thermoregulation to recuperate from the injury after a heat stroke. Until the heat intolerance test, the soldier must not train to avoid a repeat incident of heat stroke. The soldiers' ability to return to active duty is based on the results of the exam. The heat tolerance test and its criteria have been developed in the Physiology Unit throughout years of experience, and have been proved and adopted by several labs in Europe and in the United States. The criteria generally include baseline temperature and heart rate, and are based upon the physiological response of healthy men (soldiers) in the physical effort involved in the test.In recent years there is a growing trend in the IDF to integrate female soldiers in combat divisions. As a result, these females are exposed to physical efforts in various climate conditions as a part of their training, or a part of their active duty missions in the division. Therefore, the probability of an incidence of heat injuries increases among these soldiers.Research results indicate differences in the efficiency of thermoregulation mechanisms between men and women:

It has been found that in women the threshold for sweating and vasodilatation is higher than in males. Additionally, although in women the mechanism for sweating is slower, and occurs at a later period, it is found that the relative part of sweating that evaporates is higher, so that women evaporate sweat more efficiently (to make up for the lower sweat quantities compared to men). Reduced efficiency of the thermoregulation mechanisms in women is also attributed to the differences in mass, body composition (fat and muscle mass), and physical fitness between the genders. In addition, the physiological changes that occur during the different phases of the menstrual cycle can affect core temperature at rest and thermoregulation. Different reports in literature indicate a decreased thermoregulation capacity in the luteal phase of the menstrual cycle compared to the follicular phase. Apparently, thermoregulation capabilities in exercise are linked to progesterone blood levels, which are influenced by contraceptive pills and with the phase of the menstrual cycle.

There are two factors that can cause incorrect diagnosis of the level of heat tolerance in females when the specific test is interpreted based on set criteria for men. These criteria are:

1. The physiological differences between men and women
2. The differences in women based on menstrual cycle and using contraceptive pills.

Thus, there is a need to characterize and establish the normal values in a heat tolerance test for young females compared to males, and also to correspond to current menstrual cycle phase and use of contraceptive pills.

Methods:

on the first day of the research, the participants will undergo anthropometric examinations (measuring height, weight, BMI, fat content, maximum oxygen consumption). In addition, the participants will undergo a heat tolerance test protocol. The heat tolerance test will be conducted twice in every participant - once in the follicular phase of the menstrual cycle, and a second time in the luteal phase of the cycle. During the protocol, the following information will be collected from each participant: heart rate, core temperature, skin temperature in three locations (chest, arm, and leg), oxygen consumption and liquid balance.

The results of the examination will be compared to results of male participants who have previously undergone the heat tolerance test in the Unit of Military Physiology.

Contribution to IDF:

the research will allow administrating heat tolerance tests accurately and reliably to female soldiers that have been affected by heat injuries or are suspected to be heat intolerant.

ELIGIBILITY:
Inclusion Criteria:age 20-30 year, no past medical history, BMI 20-29, physically active, after completion of medical questionnaire and physical examination -

Exclusion Criteria:heart diseases, respiratory diseases,resting BP>140/90, DM, anhydrosis, skin diseases, pregnancy, breast feeding, using OC continuously, acute illness in the past two weeks.

-

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young health women
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
The physiological load in women | 1 year
  The physiological load will be mesured during a heat tolerance test (HTT) and will be compared to the physiological load during an HTT in men.

SECONDARY OUTCOMES:
Rectal temperature | 1 year
  The rectal temperature will be mesured by a rectal thermistore.
Skin temperature | 1 year
  The skin temperature will be mesured during an HTT by skin thermistores conected to 3 sites (chest, leg and arm).
Heart rate | 1 year
  The heart rate will be mesured by a polar watch.
Sweat rate | 1 year
  The sweat rate will be calculeted from the subject's weight before and after the HTT and from his water balance.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Druyan, MD, Principal Investigator — International Diabetes Federation
Locations (1):
- Sheba medical center, Ramat Gan, Israel